CLINICAL TRIAL: NCT01168245
Title: Effects of a Combined TMS Stimulation and Cognitive Training in Alzheimer Patients: a Single-center, Randomized, Double-blind, Placebo-controlled Study
Brief Title: TMS Stimulation and Cognitive Training in Alzheimer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuronix Ltd (Industry)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX-NICE-PLA02
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Alzheimer Disease; Mild to Moderate
Keywords: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Disease; Cognitive Training; Cortical Reorganization; Brain Plasticity
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NICE-System NeuroAD (Experimental): Treatment Group
  Interventions: Device: NICE-System
- Sham-TMS (Sham Comparator): Control Group
  Interventions: Device: Sham-NICE-System

INTERVENTIONS:
Device: Sham-NICE-System — sham TMS and sham cognitive training
  Other Names: NICE-System
  Arms: Sham-TMS
Device: NICE-System — TMS combined with cognitive training
  Arms: NICE-System NeuroAD

SUMMARY:
The aim of this study is to examine if combined treatment with TMS and cognitive training (CoTra) for several weeks can produce a sustained improvement in cognitive and behavioral symptomatology of mild to moderate Alzheimer's disease (AD) patients.

DETAILED DESCRIPTION:
The current available pharmaceutical treatment for Alzheimer Disease (AD) is only partially and temporary effective. Therefore, new approaches are needed. rTMS is a non-invasive technique which generates a small electric current that induces a modulation in cortical excitability. In addition, cognitive training was suggested to improve cognitive functions in Alzheimer patients.

In this study we intend to treat mild to moderate AD patients with rTMS interlaced with cognitive training (rTMS- COG).

Patients with probable AD will be treated with rTMS-COG daily for 6 weeks followed by maintenance sessions for additional 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 55-85 years
* Patients diagnosed with early or moderate stage of Alzheimer's disease, according to the DSM-IV criteria.
* MMSE score 18 to 24
* Global Dementia rating 1 or 2
* Physically acceptable for the study as confirmed by medical history and exam, clinical laboratory results and EKG
* Spouse, family member or professional caregiver agree and capable of taking care and responsibility for the participation of the patient in the study (answering questions regarding the patient's condition and assuming responsibility for medication)
* Written informed consent by both patient and legally responsible caregiver.
* Able to undergo MRI scan and EEG recordings prior to the onset of the study.
* Agreement to participate in up to 9 months the study.
* Right handed
* Hebrew or Russian as mother tongue and/or ability to read and understand the inform consent form (ICF), and the Patient Information document in Hebrew or Russian.

Exclusion Criteria:

* Severe agitation;
* Mental retardation;
* Unstable medical condition;
* Use of benzodiazepines or other hypnotics during the study and preceding two weeks;
* Pharmacological immunosuppression;
* Participation in a clinical trial with any investigational agent within two weeks prior to study enrollment;
* Alcoholism;
* History of Epileptic Seizures or Epilepsy;
* Contraindication for performing MRI scanning;
* Contraindication for receiving TMS treatment according to a TMS questionnaire;
* Clinically significant abnormal laboratory findings which have not been approved by the Principle Investigator;
* Patients treated with cholinesterase inhibitors, or memantine or ginko-biloba will be allowed to participate, if the treatment has started at least 2 months previous to recruited.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
A significant improvement and/or improvement of at least 2 points on ADAS-COG of the Treatment Group in comparison with the Placebo Group after 6 weeks of treatment. | pre-treatment, 6, and 18 weeks

SECONDARY OUTCOMES:
Safety profile: rate of device and/or procedure related adverse events. | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rabey, Prof., Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Beer Yaakov, Israel

REFERENCES:
- [Result] Rabey JM, Dobronevsky E, Aichenbaum S, Gonen O, Marton RG, Khaigrekht M. Repetitive transcranial magnetic stimulation combined with cognitive training is a safe and effective modality for the treatment of Alzheimer's disease: a randomized, double-blind study. J Neural Transm (Vienna). 2013 May;120(5):813-9. doi: 10.1007/s00702-012-0902-z. Epub 2012 Oct 18. PMID 23076723